CLINICAL TRIAL: NCT01453816
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Into the Renal Artery and Intravenously in Patients With Renal Failure
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered in Patients With Renal Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants and no longer working with off shore center
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-RF-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Renal Failure
Keywords: Renal insufficiency; kidney failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Harvesting and Isolation of Stem cells — Adipose-Derived Stem Cells (ASCs) will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered via catheter into the renal artery and intravenously.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with Renal Failure and clinical outcomes

DETAILED DESCRIPTION:
Adipose-Derived Stromal Cells (ASCs) are a novel therapy for patients suffering from Renal failure. By injecting ASCs, these regions may become populated with the ASCs, thereby potentially restoring kidney function. ASCs are a patient-derived ("autologous") cell transplantation technology that is delivered to the patient. The therapy is composed of cells derived from a patients' own adipose tissue that are isolated within approximately 1 hour and immediately delivered back to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Chronic Kidney Disease(CKD) patients of stage III, IV, or V
* Patient should be afebrile 24 hours prior to procedure.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society.

Exclusion Criteria:

* Acute Renal Failure
* Severe co-morbidities like cardiac insufficiency, congestive cardiac failure, malignancy, infection, sepsis and bed sores.
* Hemoglobin level below 6g/dl or at the discretion of the physician depending on patient's overall condition.
* Chronic kidney disease due to autoimmune aetiology, connective tissue disease, amyloidosis and storage disorders.
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for Human immunodeficiency virus (HIV), Human T-lymphotropic virus(HTLV), Hepatitis B (HBV),Hepatitis C (HCV), Cytomegalovirus (CMV) and/or syphilis will be evaluated by an expert as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg or greater than 200mmHg
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Significant clinical improvement in serum creatinine and urine output (improvement in measured Glomerular Filtration Rate(GFR) by 50%) | 3 months
  Compared to baseline
number of participants with adverse events | 1 week
Significant clinical improvement in serum creatinine and urine output (improvement in measured Glomerular Filtration Rate(GFR) by 50%) at 6 months | 6 months
number of participants with adverse events | 2 weeks
number of participants with adverse events | 4 weeks

SECONDARY OUTCOMES:
Improvement in renal biopsy measured by the reduction of scarring etc as compared to baseline | 3 months
Improvement in renal biopsy measured by the reduction of scarring etc as compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rigoberto Pallares, MD, Principal Investigator — Instituto de Medicina Regenerativa
Locations (1):
- Hospital Angeles, Tijuana, Estado de Baja California, Mexico